CLINICAL TRIAL: NCT02591810
Title: Comparison of Treatment Options for Acute Distal Radioulnar Joint Instability: A Prospective Randomized Control Trial
Brief Title: Treatment Options for Acute Distal Radioulnar Joint Instability
Acronym: DRUJ
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Orlando Health, Inc. (Other)
Responsible Party: Principal Investigator, Brett Lewellyn, Orthopedic surgeon, Hand specialist, Orlando Health, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15.041.04
Record Dates: First submitted 2015-07-22; First posted 2015-10-30 (Estimated); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Wrist Injuries
MeSH Terms: conditions — Wrist Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Serial Casting (Active Comparator): Participants will receive the intervention of the placement of serial casting/splinting for the injured wrist. This is not a surgical intervention.
  Interventions: Procedure: Serial casting/splinting
- Kirschner wires (Active Comparator): Participants will receive the intervention of percutaneous fixation with Kirschner wires for the injured wrist. This will be performed surgically.
  Interventions: Procedure: Percutaneous fixation
- Foveal repair (Active Comparator): Participants will receive the intervention of open anatomic foveal repair of the ligaments of the injured wrist. This is a surgical intervention.
  Interventions: Procedure: Foveal repair

INTERVENTIONS:
Procedure: Serial casting/splinting — Serial Casting involves applying and removing a series of lightweight casts made of fiberglass. The wrist is monitored as healing occurs.
  Arms: Serial Casting
Procedure: Percutaneous fixation — Injury is treated by the percutaneous placement of Kirschner wires to promote healing. This is an invasive procedure, involving the placement of Kirschner wires to stabilize the wrist.
  Arms: Kirschner wires
Procedure: Foveal repair — Injury is treated by open anatomic foveal repair of the ligaments. This is a surgical procedure.
  Arms: Foveal repair

SUMMARY:
This prospective randomized control trial (PRCT) aims to compare the outcome of three treatments for acute distal radioulnar joint (DRUJ) injury with instability with or without concomitant distal radius fractures: serial splinting/casting with the hand and wrist in the most stable position for DRUJ reduction vs percutaneous DRUJ fixation with Kirschner wires vs open anatomic foveal repair of Triangular fibrocartilage complex (TFCC ) ligaments.

DETAILED DESCRIPTION:
This is a prospective randomized control trial comparing three methods of treatment for acute DRUJ instability with or without concomitant distal radius fracture. Upon determination of residual DRUJ instability either preoperatively or intraoperatively after distal radius fracture fixation, patients will be randomized into one of the three treatment arms of the study: nonoperative treatment with immobilization, percutaneous DRUJ fixation with Kirschner wires, and open anatomic foveal repair of Triangular fibrocartilage complex TFCC ligaments with suture. Those patients undergoing Kirschner wire fixation will have their pins pulled in the clinic setting six weeks postoperatively. Outcomes will be assessed at follow up visits using the subjective and objective measures and clinical assistants will be blinded as to the treatment type. Physician-based assessment of functional outcome with be assessed using the Disability of the Arm, Shoulder and Hand (DASH) score and Mayo Wrist scores, as well as independent assessment of DRUJ instability, ROM, and grip strength. Patient-based assessment will include visual analog pain scores as well as satisfaction questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Patients treated at Orlando Regional Medical Center,
2. 18 years or older,
3. Have an acute (less than 4 week old) injury with instability of the DRUJ.

Exclusion Criteria:

1. Younger than 18 years old,
2. Patients with an injury over 4 weeks old,
3. Previous history of ipsilateral upper extremity trauma,
4. Functional deficit,
5. Those who are unable to complete postoperative assessments. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11-05 (Actual); Primary Completion 2016-11-05 (Actual); Study Completion 2016-11-09 (Actual)

PRIMARY OUTCOMES:
Evaluation and assessment of DASH scores. | Up to 5 years.
  To compare the outcomes of the three treatment arms for acute DRUJ instability by assessment with the Disabilities of the Arm, Shoulder, and Hand (DASH) Score.

SECONDARY OUTCOMES:
Visual Analog Pain scale | Up to 5 years.
  Patient will be asked to describe level on pain on a 10cm scale, in 1 cm increments, from 0 to 10. 0 equals no pain, 10 equals the worst pain.

OTHER OUTCOMES:
Mayo wrist assessment scores | Up to 5 years
  Patients will be asked to describe their pain intensity, range of motion, grip strength and functional status.
Patient satisfaction | Up to 5 years
  Patients will be asked to describe on a scale from 1 to 10 how satisfied they are with their surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Tara Roberts, BS, Study Chair — Orlando Health